CLINICAL TRIAL: NCT06391606
Title: Effect of Coenzyme Q10 on Physical Performance in Elderly Patients With Statin-associated Asthenia: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: CoQ10 in Statin-associated Asthenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Prof. Dr., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QELD_Stat_2017
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hypercholesterolemia; Physical Performance
Keywords: Statin; Asthenia; Coenzyme Q10
MeSH Terms: conditions — Hypercholesterolemia; Asthenia | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 (Active Comparator): 2 pills of 150 mg CoQ10 phytosome (i.e. 300 mg CoQ10 phytosome per day)
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): 2 pills of placebo per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 2 pills/day of 150 mg CoQ10 phytosome (i.e. 300 mg CoQ10 phytosome per day)
  Arms: Coenzyme Q10
Other: Placebo — 2 pills/day
  Arms: Placebo

SUMMARY:
This was a double-blind, randomized, placebo-controlled clinical study aiming to assess the effects of supplementation with CoQ10 phytosome on physical performance in older adults with self-reported statin-associated asthenia.

ELIGIBILITY:
Inclusion criteria:

* 65-80 years of age
* treatment for >6 months with statin monotherapy (i.e. enrolled individuals were asked to be on the same statin at the same dosage for >6 months)
* statin-associated asthenia for >3 months

Exclusion criteria:

* serious or disabling diseases (e.g. severe organ failure, malignancy or dementia)
* orthopedic disorders, myopathies and any other acute or chronic disease that could significantly affect the individual's perception of asthenia
* obesity (body mass index (BMI)> 30 Kg/m2)
* known gastrointestinal disorders potentially affecting the absorption of CoQ10

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Effect on handgrip strength | 8 weeks
  We evaluated the effect on handgrip strength after 8 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
  A hand-held dynamometer was used to assess handgrip strength. Measurements were assessed according to the International standard protocols, and obtained after participants performed one familiarization trial with both hands.

SECONDARY OUTCOMES:
Effect on handgrip strength | 4 weeks
  We evaluated the effect on handgrip strength after 4 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
  A hand-held dynamometer was used to assess handgrip strength. Measurements were assessed according to the International standard protocols, and obtained after participants performed one familiarization trial with both hands.
Effect on statin-associated asthenia | 4 weeks
  We evaluated the effect on asthenia after 4 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
  Asthenia was assessed on a 10-point visual analogue scale (VAS), considering 0= absence of asthenia and 10= extreme asthenia.
Effect on statin-associated asthenia | 8 weeks
  We evaluated the effect on asthenia after 8 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
  Asthenia was assessed on a 10-point visual analogue scale (VAS), considering 0= absence of asthenia and 10= extreme asthenia.
Effect on 1-min sit-to-stand repetitions | 4 weeks
  We evaluated the effect on 1-min sit-to-stand repetitions after 4 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
Effect on 1-min sit-to-stand repetitions | 8 weeks
  We evaluated the effect on 1-min sit-to-stand repetitions after 8 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
Effect on 2-minute step test | 4 weeks
  We evaluated the effect on 2-minute step test after 4 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.
Effect on 2-minute step test | 8 weeks
  We evaluated the effect on 2-minute step test after 8 weeks of dietary supplementation with CoQ10 phytosome compared to either baseline and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, PhD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No